CLINICAL TRIAL: NCT06213181
Title: Effects of an Intervention Based on Mindfulness on the Physical and Mental Condition in People Over 65 Years of Age With Chronic Musculoskeletal Pain
Brief Title: Mindfulness on Physical and Mental Condition in Older Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: -University_of_Jaén
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: To assign participants to the control and intervention groups, random sampling will be carried out using sealed and completely opaque envelopes. It will be carried out by a researcher who will not intervene in the different phases of the intervention: neither in the initial phase nor in the subsequent evaluation phase. Therefore, the rest of the researchers will not know to which group each participant who has been included in the study has been assigned.The assignment will be communicated using sealed and totally opaque envelopes. The analysis of the results will be carried out by a researcher unrelated to the group assignment and the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants assigned to this group will receive general advice about the positive effects of regular physical activity. They will be given a guide of physical exercise recommendations, according to the World Health Organization for people over 65 years of age.
- Mindfulness intervention (Experimental): Participants assigned to this group will receive a mindfulness-based intervention for eight weeks with a weekly session lasting two hours per session. It is an experimental and interactive program that includes conscious movements, meditation, practical activities on attention in the present moment and the search for strategies to face complex situations from the collective and individual level. Participants will carry out daily practices at home during the week with the resources shared in each session.
  Interventions: Other: Mindfulness intervention

INTERVENTIONS:
Other: Mindfulness intervention — It consists of 8 weekly sessions with a duration of 2 hours each. A variety of mindfulness practices including mindful movement will be introduced in all sessions. Participants will approach meditation as something natural and everyday, with the possibility of directing attention in all the moments and activities of daily life. Body scanning practices and conscious breathing will also be included. We will work in the group, with reflections and readings, as well as carrying out meditation and mindfulness practices, during the week, so that they can be carried out in the daily life of each participant. The intervention based on mindfulness will focus on the areas of well-being and personal skills such as attention, communication, emotional regulation and decision making.
  Arms: Mindfulness intervention

SUMMARY:
This research corresponds to an experimental study, a randomized controlled clinical trial in people over 65 years of age, distributed into two groups: the experimental group will receive a program that will consist of an eight-week mindfulness-based intervention; and the control group that will only receive general recommendations about the benefits of physical exercise. Measurements will be carried out at the beginning of the intervention and immediately after its completion.

ELIGIBILITY:
Inclusion Criteria:

* The study participants are men and women over 65 years of age residing in the city of Jaén (Spain).
* People with pain with more than 3 months of evolution.
* Participants must have completed the informed consent.

Exclusion Criteria:

* That they do not voluntarily accept to participate in the study and that they are able to understand the instructions and follow the instructions of the intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
SF-12 (reduced version of The Health Survey Short Form-36) | Up to twelve weeks
  Used extensively for assessing health-related quality of life. The results are values between 0 and 100. Optimal health is represented by scores of 100 and very poor health would equal 0.
Numeric Rating Scale (NRS) | Up to twelve weeks
  Patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
FSS (Fatigue Severity Scale) | Up to twelve weeks
  A self-report scale describing the severity of fatigue and the impact of fatigue on activities of daily living. The test is made up of 9 items with 7 response possibilities, so that 1 and 7 correspond to the minimum and maximum severity respectively. The total score corresponds to the sum of all the items with a total score range that goes from 9 to 63.
PSQI (Pittsburgh Sleep Quality Index) | Up to twelve weeks
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result. Higher scores indicate poorer sleep. It contains a total of 19 questions, grouped into 10 questions. The 19 questions are combined to form seven areas with their corresponding score, each of which shows a range between 0 and 3 points. In all cases, a score of "0" indicates ease, while a score of 3 indicates severe difficulty, within their respective area. The scores of the seven areas are finally added to give an overall score, which ranges between 0 and 21 points. "0" indicates ease of sleeping and "21" severe difficulty in all areas.
PSS (Perceived Stress Scale) | Up to twelve weeks
  It consists of 14 items with a five-point scale response format (0 = never, 1 = almost never, 2 = occasionally, 3 = often, 4 = very often). The total score of the PSS is obtained by reversing the scores of items 4, 5, 6, 7, 9, 10 and 13 (in the following sense: 0=4, 1=3, 2=2, 3=1 and 4 =0) and then adding the 14 items. The direct score obtained indicates that a higher score corresponds to a higher level of perceived stress.
Chair stand test | Up to twelve weeks
  Evaluate the strength of the lower body. The total number of times you "get up and sit down" in the chair for 30" is counted. If at the end of the exercise the participant has completed half or more of the movement (standing up and sitting down), it will be counted as complete.
TUG test (Timed Up and Go test) | Up to twelve weeks
  Is a simple test used to assess a person's mobility and physical function.
Tinetti scale | Up to twelve weeks
  It is used to determine early the risk of falling in an elderly person during the year following its application. The result of both sections will be added, so that a score of less than 19 points will imply a high risk of falls, a score of 19 to 24 will reflect medium risk of falls and a score of 25 to 28 will indicate low risk of falls.
HADS (The Hospital Anxiety And Depression) | Up to twelve weeks
  A reliable, valid and practical screening tool for identifying and quantifying anxiety and/or depression in non-patients. The test contains 14 items with a score from 0 to 3, of which 7 items refer to depression and 7 to anxiety. The total score is 0-21, where a higher score corresponds to worse symptoms of anxiety and depression.
Arm curl test | Up to twelve weeks
  Evaluate upper body strength. The total number of times the arm is "flexed and extended" during 30" is counted. If at the end of the exercise the participant has completed half or more of the movement (flexion and extension of the arm), it will be counted as complete.
Back scratch test | Up to twelve weeks
  Evaluate the flexibility of the upper body (mainly the shoulders). The participant will make two attempts with the best side before starting the test and it will be noted on the record sheet by putting a circle in the best of them.
Chair-sit and reach-test | Up to twelve weeks
  Evaluate the flexibility of the lower body (mainly biceps femoris). The participant will perform two attempts with the preferred leg and the examiner will record the two results by circling the best of them on the recording sheet. The distance is measured from the tips of the fingers of the hands to the top of the shoe. Touching the toe of the shoe will score "Zero". If the fingers of the hands do not reach the foot, the distance will be measured in negative values (-). If the fingers of the hands exceed the foot, the distance is recorded in positive values (+).
Brief Pain Questionnaire (CBD) | Up to twelve weeks
  It is a multidimensional pain assessment instrument that provides information on the intensity of pain and its interference with patients' daily activities. Also assess the description, location of the pain and the level of relief provided by the treatment.

SECONDARY OUTCOMES:
BMI (Body Mass Index) | Up to twelve weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat
Waist circumference | Up to twelve weeks
  Is used to assess central fat distribution and degree of abdominal obesity
Hip circumference | Up to twelve weeks
  It is measured at the level of the maximum prominence of the buttocks.

CONTACTS AND LOCATIONS:
Locations (1):
- Municipal social services center "el boulevard", Jaén, Spain